CLINICAL TRIAL: NCT05679726
Title: The Effect of Foot Reflexology on Stress, Fatigue and Low Back Pain in Intensive Care Nurses
Brief Title: The Effect of Foot Reflexology in Intensive Care Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Ayse Gul Parlak, assistant proffessor, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: kafkasU-80576354
Record Dates: First submitted 2023-01-02; First posted 2023-01-11 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Fatigue; Pain; Stress; Nurse
MeSH Terms: conditions — Fatigue; Pain | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (reflexology group) (Experimental): The group in which reflexology massage (foot massage) was applied once a week for 20 minutes (10 minutes on each foot) for a total of 4 weeks, and the pain scale and fatigue and stress level were measured once a week at the beginning of the study and at the end of the study 4 weeks later.
  Interventions: Behavioral: massage
- Control group (No Intervention): Pain scale once a week for 4 weeks without any application, and fatigue and stress level at the beginning of the study and at the end of the study after 4 weeks were measured in the group.

INTERVENTIONS:
Behavioral: massage — reflexology foot massage
  Arms: Intervention group (reflexology group)

SUMMARY:
This study was planned as a randomized controlled experimental research design to examine the effect of foot reflexology applied to nurses working in the intensive care unit on stress, fatigue and low back pain.

DETAILED DESCRIPTION:
The universe of the research consisted of a total of 90 nurses working in a university and a public hospital in a city. Among the nurses, those who meet the criteria for inclusion in the study will form the sample. Assignment to the intervention and control group will be determined in the computer environment using a simple randomization method (www.randomizer.org/). The number of samples was determined using power analysis. It was decided to recruit a total of 42 nurses, 21 for each group.

ELIGIBILITY:
Inclusion Criteria:

* -Intensive care unit nurse
* Those aged 18 to 65 years
* Working in intensive care for at least 6 months
* Back pain for at least 3 months
* Not pregnant, non-breastfeeding
* Having a regular menstrual cycle
* Vascular disease and foot fracture, wound, scar, skin damage etc. no situation
* Volunteered to participate in the research
* Not using antidepressants, sleeping pills, etc.

Exclusion Criteria:

* Working in intensive care for less than 6 months
* No chronic low back pain
* Pregnant, lactating
* Do not have a regular menstrual cycle
* Vascular disease and foot fracture, wound, scar, skin damage etc. situation found
* Using antidepressants, sleeping pills, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
pain severity | pre test
  measurement of nurses' low back pain severity score
  A Visual Analogue Scale (VAS) is one of the pain rating scales. VAS pain score is evaluated as "painless" (score=0) and "worst pain" (score=10).
  score <3 mild pain, 3-6 mild-to-moderate pain, and >6 moderate-to-severe pain
fatique | pre test
  The fatigue severity scale There are 9 questions in the scale and each question consists of 7 points. An increase in the scale score indicates an increase in the level of fatigue. The scale determines the fatigue status of individuals in the last 1 month. Questions are scored as I totally disagree (1)- I totally agree. If the average score is 5 and above, it is considered as "fatigue".
stress | pre test
  Perceived Stress Scale ; There are 14 items in the scale, which was developed as a five-point Likert-type rating scale. The scale consists of "never (0), almost never" (1), "sometimes" (2), "often" (3) "very often" (4). The lowest and highest scores a participant can obtain from this scale are 0 and 56, respectively.

SECONDARY OUTCOMES:
pain severity | post test(at the end of the 4th week)
  measurement of nurses' low back pain severity score
  A Visual Analogue Scale (VAS) is one of the pain rating scales. VAS pain score is evaluated as "painless" (score=0) and "worst pain" (score=10).
  score <3 mild pain, 3-6 mild-to-moderate pain, and >6 moderate-to-severe pain
fatique | post test (at the end of the 4th week)
  The fatigue severity scale There are 9 questions in the scale and each question consists of 7 points. An increase in the scale score indicates an increase in the level of fatigue. The scale determines the fatigue status of individuals in the last 1 month. Questions are scored as I totally disagree (1)- I totally agree. If the average score is 5 and above, it is considered as "fatigue".
stress | post test(at the end of the 4th week)
  Perceived Stress Scale ; There are 14 items in the scale, which was developed as a five-point Likert-type rating scale. The scale consists of "never (0), almost never" (1), "sometimes" (2), "often" (3) "very often" (4). The lowest and highest scores a participant can obtain from this scale are 0 and 56, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Gül Parlak, PhD, Principal Investigator — Kafkas University
Locations (1):
- Ayşe Gül Parlak, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No